CLINICAL TRIAL: NCT03270280
Title: Comparison of Salivary Interleukin-1β and Matrix Metalloproteinase-8 Levels in Individuals With Chronic Periodontitis Before and After Treatment With Nigella Sativa (Kalonji) Oil
Brief Title: Comparison of Salivary Interleukin-1β and Matrix Metalloproteinase-8 Levels in Individuals With Chronic Periodontitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Dr. Ghazala Hassan, Research Scholar, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: UniversityHSL
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Chronic Periodontitis
Keywords: Chronic Periodontitis; Phytomedicines; Nigella sativa
MeSH Terms: conditions — Chronic Periodontitis | interventions — Nigella sativa oil; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Healthy Individuals with Chronic Periodontitis Only
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal Saline (Placebo Comparator): The group contains healthy individuals with chronic periodontitis who will receive Normal Saline as placebo
  Interventions: Drug: Normal saline
- Nigella Sativa (Experimental): The group contains healthy individuals with chronic periodontitis who will receive Nigella sativa Oil as intervention
  Interventions: Drug: Nigella Sativa Oil

INTERVENTIONS:
Drug: Nigella Sativa Oil — The individuals will apply 55 drops of Nigella sativa Oil on gingivae twice daily for two weeks
  Other Names: Black seed Oil
  Arms: Nigella Sativa
Drug: Normal saline — The individuals will apply 55 drops of Normal saline on gingivae twice daily for two weeks
  Other Names: Saline
  Arms: Normal Saline

SUMMARY:
Periodontitis is an infectious inflammatory disease affecting the periodontal tissue (Gingivae, alveolar bone, periodontal ligament and cementum). Chronic Periodontitis is considered to be the most prevalent disease after dental caries which is linked to increased levels of C- reactive protein, interleukins and matrix metallo-proteinases. Interleukin- 1β and Matrix metalloproteinase-8 have been shown to be robust markers of inflammatory cascade of chronic periodontitis.Various treatment modalities including scaling and root planing, toothpastes and chlorhexidine based mouthwashes have been are known to be associated with various side effects like teeth staining, altered taste sensation, mucosal burning. Hence,the use of natural medicaments could provide a better alternative because of their fewer side effects and cost effectiveness.

DETAILED DESCRIPTION:
Periodontal disease is one of the most common diseases in humans and is responsible for most of the tooth loss in adults. World health Organisation report of 2005 described that the global problem persisted with the worldwide oral diseases such as dental caries, periodontal disease, tooth loss, oral mucosal lesions and oro-pharyngeal cancer. According to a local study the prevalence of periodontitis is found to be more in males of older age group and more in rural areas owing to the lack of awareness of importance of oral hygiene.

Apart from various conventional treatment option for periodontitis a number of herbal medicinal intervention have been used for its treatment. Plant extracts and herbs that have been used previously used for periodontal therapy include Salvadora persica, Arnica Montana and Hamamelis virginiana which have been shown to exhibit antibacterial activity against periodonto-pathic bacteria. Phytomedicines (Medicines derived from herbal plants) like indian gum arabic, aloe vera, nim, carvacrol, garlic, wild coffee and propolis resin have been used in dentistry as anti-inflammatory, antibiotics, analgesic and hypnotic agents. Propolis resin, guava and triphala have been also been used for the treatment of periodontitis

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy individual
* Individuals diagnosed with chronic periodontitis according to the WHO criteria.
* Age 19 to 40 years.

Exclusion Criteria:

* Patients with gingivitis only.
* Patients using tobacco products and alcohol.
* Underlying systemic pathology such as diabetes mellitus, cardiovascular disease, arthritis etc.
* Oral mucosal pre-neoplastic lesions (leukoplakia, erthroplakia, lichen planus) and oral carcinomas.
* Obese patients.
* Pregnant females.
* Xerostomia.
* Previous history of radiotherapy or chemotherapy.
* Positive history of oral prophylactic procedures (mouthwashes and antibiotics).
* Positive history of any periodontal treatment during last 6 months.
* Positive antibiotic therapy history within last month of study.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-09-11 (Estimated); Primary Completion 2018-03-11 (Estimated); Study Completion 2018-04-11 (Estimated)

PRIMARY OUTCOMES:
Levels of IL 1-Beta and MMP-8 | 2 weeks
  These inflammatory marker will be measured in patients saliva again after 2 weeks. There will be reduction in their levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ghazala Hassan, MPhil, Principal Investigator — Research Scholar
Locations (1):
- Fatima Memorial Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data sharing will be considered after the completion of studies

REFERENCES:
- [Background] Zadik Y, Bechor R, Galor S, Levin L. Periodontal disease might be associated even with impaired fasting glucose. Br Dent J. 2010 May 22;208(10):E20. doi: 10.1038/sj.bdj.2010.291. Epub 2010 Mar 26. PMID 20339371
- [Background] Gupta N, Gupta ND, Gupta A, Khan S, Bansal N. Role of salivary matrix metalloproteinase-8 (MMP-8) in chronic periodontitis diagnosis. Front Med. 2015 Mar;9(1):72-6. doi: 10.1007/s11684-014-0347-x. Epub 2014 Aug 6. PMID 25098434